CLINICAL TRIAL: NCT04462796
Title: The Effect of Magnesium Citrate Supplementation in Patients With Restless Legs Syndrome (RLS) - An Open Label, Prospective, Non Placebo Controlled Pilot Study
Brief Title: The Effect of Magnesium Citrate Supplementation in Restless Legs Syndrome (RLS)
Acronym: RLS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: OSF Healthcare System (Other)
Responsible Party: Principal Investigator, Sasikanth Gorantla, Principal Investigator, OSF Healthcare System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1567451
Record Dates: First submitted 2020-07-05; First posted 2020-07-08 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Restless Legs Syndrome
Keywords: RLS, Magnesium Citrate, Magnesium
MeSH Terms: conditions — Restless Legs Syndrome | interventions — magnesium citrate

STUDY DESIGN:
Intervention Model Description: Pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Magnesium Citrate (Experimental): Magnesium Citrate given orally taken once daily for 8 weeks
  Interventions: Dietary Supplement: Magnesium Citrate

INTERVENTIONS:
Dietary Supplement: Magnesium Citrate — Magnesium Citrate 200 mg daily

SUMMARY:
The expected results of this study will have a significant impact on the treatment of RLS/WED patients. Magnesium supplementation (if proven to be beneficial) can be utilized as an inexpensive, safer, biologically plausible alternative to dopamine agonists and α2δ calcium-channel ligands.

DETAILED DESCRIPTION:
This is an open-label, prospective, non-placebo controlled pilot study. 15 subjects with a diagnosis of restless legs syndrome (ICSD-3 diagnostic criteria) will be recruited from OSF Healthcare Saint Francis Medical Center sleep center and Illinois Neurological Institute. RLS/WED patients who meet inclusion and exclusion criteria during the initial clinic visit will be offered study participation. Standard treatment options will be discussed prior to the enrollment. Patients will be reassured that not participating in the study will not affect the future care they receive at OSF HealthCare. The potential risks and benefits of the study will be provided and, if the patient is interested, informed consent will be obtained. If the subject withdraws consent or does not finish both pre and post evaluation, we will replace the subject with another new recruit. The subject will come to the clinic for 2 visits, a pre-magnesium visit and a post-magnesium visit. Following the completion of the pre-magnesium visit, the subject will be given 200 mg elemental magnesium daily (will be instructed to take with food at dinner) for 8 weeks. Both Visits the following study procedures will be performed: magnesium level, (International Restless Legs Syndrome) IRLS scale, Kohnen Restless Legs Syndrome Quality of Life Instrument (KRLS-QOL) scale and (Multiple Suggested Immobilization (MSI) test. The post magnesium visit will be schedule at the completion of the 8 week dose of magnesium.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 89.
2. Treatment naïve patients (who are not taking RLS medications for at least 1 year) without coexisting untreated OSA.
3. Diagnosed with RLS based on ICSD -3 criteria
4. INI OSF Sleep medicine outpatient clinic patients.
5. Patients with the ability to provide informed consent.

Exclusion Criteria:

1. Patients who are currently taking magnesium supplements or took magnesium supplements in the last 3 months.
2. Patients not on a stable dosage of medications ( patients requiring dosage changes) that can cause PLMs or worsen RLS will be excluded ( medications include antidepressants such as SSRIs, SNRIs and TCAs and Antihistamines such as Benadryl and Allegra, etc)
3. Patients with a history of chronic kidney disease or end-stage renal disease on Hemodialysis
4. Patients with known allergies to magnesium citrate
5. Patients with congestive heart failure with an ejection fraction less than 40%, bradycardia with a resting heart rate below 60 and systolic blood pressure less than 90 mm of Hg.
6. Patients with diarrhea
7. Patients on gabapentin or pregabalin for pain syndromes
8. Pregnancy. (Absence of pregnancy will be determined via subject self-reporting only. Subject self-reporting of the absence of pregnancy is sufficient screening because the dosage of Magnesium supplement that subjects will be consuming during the study is well below the NIH Tolerable Upper Intake Levels for pregnancy [see "Dietary Recommendations" below], and has been shown to cause no fetal abnormalities or pregnancy complications at the dosage patients will consume for the study. Subjects will be encouraged to practice appropriate measures to avoid pregnancy throughout the entirety of their study participation).

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2020-07-10 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Subjective Improvement of Restless Legs Symptoms measured by the International Restless Legs Syndrome Scale (IRLS) | Completion of Study participation at 8 weeks
  International Restless Leg Syndrome Scale. (IRLS) is a 10 question scale that subjects rate on a scale of 0-4; RLS can be classified as mild, moderate, severe and very severe, if the score is 0-10 (mild), 11-20 (moderate), 21-30 (severe) or 31-40 (very severe) respectively. The lower score reflects less symptom burden. Minimum score is 0 with a Maximum of 40.
Subjective Improvement of Restless Legs Symptoms measured by the Kohnen Kohnen Restless Legs Syndrome Quality of Life Instrument (KRLS QOL) | Completion of Study participation at 8 weeks
  Kohnen Restless Legs Syndrome Quality of Life instrument (KRLS QOL) is a self-administered validated patient-reported outcome measure with 12 questions that assess the quality of life in RLS patients. Scores range from 0-60.The lower score represents less impact of RLS symptoms on quality of life.
Objective Improvement of Restless Legs Symptoms: Multiple Suggested Immobilization test (MSI) Score | Completion of Study participation at 8 weeks
  Reduction in Multiple Suggested Immobilization test (MSI) discomfort Scores, range: 0-10, with a maximum total sum of 60 per hour. Three 1 hour trials will be conducted. Periodic limb movements during wakefulness will also be measured. Periodic limb movement index (PMLI) reflects periodic limb movements per hour. PMLI value of 0 indicates absence of limb movements and higher scores are often seen in patients with severe RLS
Correlation of magnesium levels with Kohnen Restless Legs Syndrome Quality of Life Instrument (KRLS) and Multiple Suggested Immobilization test (MSI) scores | Completion of Study participation at 8 weeks
  Assessment of Magnesium level, lab value will be assess. Normal values range from 1.6 - 2.6 mg/dl. The rationale of measuring serum magnesium level is to analyze whether serum magnesium levels correlate with other subjective and objective RLS outcome measures

CONTACTS AND LOCATIONS:
Overall Officials: Sasikanth Gorantla, MD, Principal Investigator — OSF Healthcare Saint Francis Medical Center
Locations (1):
- OSF Healthcare Illinois Neurological Institute, Peoria, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided
Plan to share an abstract and data analysis results.

REFERENCES:
- [Background] Pratt DP. Restless Legs Syndrome/Willis-Ekbom Disease and Periodic Limb Movements: A Comprehensive Review of Epidemiology, Pathophysiology, Diagnosis and Treatment Considerations. Curr Rheumatol Rev. 2016;12(2):91-112. doi: 10.2174/1573403x12666160223120340. PMID 26902775
- [Background] Montplaisir J, Boucher S, Poirier G, Lavigne G, Lapierre O, Lesperance P. Clinical, polysomnographic, and genetic characteristics of restless legs syndrome: a study of 133 patients diagnosed with new standard criteria. Mov Disord. 1997 Jan;12(1):61-5. doi: 10.1002/mds.870120111. PMID 8990055
- [Background] Coleman RM, Miles LE, Guilleminault CC, Zarcone VP Jr, van den Hoed J, Dement WC. Sleep-wake disorders in the elderly: polysomnographic analysis. J Am Geriatr Soc. 1981 Jul;29(7):289-96. doi: 10.1111/j.1532-5415.1981.tb01267.x. PMID 7240617
- [Background] Scofield H, Roth T, Drake C. Periodic limb movements during sleep: population prevalence, clinical correlates, and racial differences. Sleep. 2008 Sep;31(9):1221-7. PMID 18788647
- [Background] Garcia-Borreguero D, Guitart X, Garcia Malo C, Cano-Pumarega I, Granizo JJ, Ferre S. Treatment of restless legs syndrome/Willis-Ekbom disease with the non-selective ENT1/ENT2 inhibitor dipyridamole: testing the adenosine hypothesis. Sleep Med. 2018 May;45:94-97. doi: 10.1016/j.sleep.2018.02.002. Epub 2018 Feb 24. PMID 29680437
- [Background] Leu-Semenescu S, Petiau C, Charley Monaca C, Dauvilliers Y. French consensus: Augmentation syndrome in restless legs syndrome. Rev Neurol (Paris). 2018 Sep-Oct;174(7-8):532-539. doi: 10.1016/j.neurol.2018.06.004. Epub 2018 Jul 25. PMID 30055794
- [Background] Ito E, Inoue Y. [The International Classification of Sleep Disorders, third edition. American Academy of Sleep Medicine. Includes bibliographies and index]. Nihon Rinsho. 2015 Jun;73(6):916-23. Japanese. PMID 26065120
- [Background] Ferini-Strambi L, Aarskog D, Partinen M, Chaudhuri KR, Sohr M, Verri D, Albrecht S. Effect of pramipexole on RLS symptoms and sleep: a randomized, double-blind, placebo-controlled trial. Sleep Med. 2008 Dec;9(8):874-81. doi: 10.1016/j.sleep.2008.09.001. Epub 2008 Oct 25. PMID 18952497
- [Background] Giorgi L, Asgharian A, Hunter B. Ropinirole in patients with restless legs syndrome and baseline IRLS total scores >/= 24: efficacy and tolerability in a 26-week, double-blind, parallel-group, placebo-controlled study followed by a 40-week open-label extension. Clin Ther. 2013 Sep;35(9):1321-36. doi: 10.1016/j.clinthera.2013.06.016. Epub 2013 Aug 9. PMID 23938061
- [Background] Walters AS, LeBrocq C, Dhar A, Hening W, Rosen R, Allen RP, Trenkwalder C; International Restless Legs Syndrome Study Group. Validation of the International Restless Legs Syndrome Study Group rating scale for restless legs syndrome. Sleep Med. 2003 Mar;4(2):121-32. doi: 10.1016/s1389-9457(02)00258-7. PMID 14592342
- [Background] Abetz L, Arbuckle R, Allen RP, Garcia-Borreguero D, Hening W, Walters AS, Mavraki E, Kirsch JM. The reliability, validity and responsiveness of the International Restless Legs Syndrome Study Group rating scale and subscales in a clinical-trial setting. Sleep Med. 2006 Jun;7(4):340-9. doi: 10.1016/j.sleep.2005.12.011. Epub 2006 May 19. PMID 16713344
- [Background] Kohnen R, Martinez-Martin P, Benes H, Trenkwalder C, Hogl B, Dunkl E, Walters AS. Validation of the Kohnen Restless Legs Syndrome-Quality of Life instrument. Sleep Med. 2016 Aug;24:10-17. doi: 10.1016/j.sleep.2016.04.019. Epub 2016 Aug 3. PMID 27810174
- [Background] Sforza E, Johannes M, Claudio B. The PAM-RL ambulatory device for detection of periodic leg movements: a validation study. Sleep Med. 2005 Sep;6(5):407-13. doi: 10.1016/j.sleep.2005.01.004. Epub 2005 Apr 1. PMID 16139771
- [Background] Garcia-Borreguero D, Kohnen R, Boothby L, Tzonova D, Larrosa O, Dunkl E. Validation of the Multiple Suggested Immobilization Test: A Test for the Assessment of Severity of Restless Legs Syndrome (Willis-Ekbom Disease). Sleep. 2013 Jul 1;36(7):1101-1109. doi: 10.5665/sleep.2820. PMID 23814348
- [Background] De Cock VC, Bayard S, Yu H, Grini M, Carlander B, Postuma R, Charif M, Dauvilliers Y. Suggested immobilization test for diagnosis of restless legs syndrome in Parkinson's disease. Mov Disord. 2012 May;27(6):743-9. doi: 10.1002/mds.24969. Epub 2012 Mar 21. PMID 22437899
- [Background] Marshall NS, Serinel Y, Killick R, Child JM, Raisin I, Berry CM, Lallukka T, Wassing R, Lee RW, Ratnavadivel R, Vedam H, Grunstein R, Wong KK, Hoyos CM, Cayanan EA, Comas M, Chapman JL, Yee BJ. Magnesium supplementation for the treatment of restless legs syndrome and periodic limb movement disorder: A systematic review. Sleep Med Rev. 2019 Dec;48:101218. doi: 10.1016/j.smrv.2019.101218. Epub 2019 Oct 16. PMID 31678660
- [Background] Hornyak M, Voderholzer U, Hohagen F, Berger M, Riemann D. Magnesium therapy for periodic leg movements-related insomnia and restless legs syndrome: an open pilot study. Sleep. 1998 Aug 1;21(5):501-5. doi: 10.1093/sleep/21.5.501. PMID 9703590
- [Background] Bartell S, Zallek S. Intravenous magnesium sulfate may relieve restless legs syndrome in pregnancy. J Clin Sleep Med. 2006 Apr 15;2(2):187-8. PMID 17557494
- [Background] Institute of Medicine (US) Standing Committee on the Scientific Evaluation of Dietary Reference Intakes. Dietary Reference Intakes for Calcium, Phosphorus, Magnesium, Vitamin D, and Fluoride. Washington (DC): National Academies Press (US); 1997. Available from http://www.ncbi.nlm.nih.gov/books/NBK109825/ PMID 23115811
- [Background] [The unveiling ceremony of the monument of the Unknown Nurse]. Noseleutike. 1992 Jan-Mar;31(139):19-23. No abstract available. Greek, Modern. PMID 1596323
- [Background] Coudray C, Rambeau M, Feillet-Coudray C, Gueux E, Tressol JC, Mazur A, Rayssiguier Y. Study of magnesium bioavailability from ten organic and inorganic Mg salts in Mg-depleted rats using a stable isotope approach. Magnes Res. 2005 Dec;18(4):215-23. PMID 16548135
- [Background] Lowenstein FW, Stanton MF. Serum magnesium levels in the United States, 1971-1974. J Am Coll Nutr. 1986;5(4):399-414. doi: 10.1080/07315724.1986.10720143. PMID 3771947
- [Background] Michaud M, Poirier G, Lavigne G, Montplaisir J. Restless Legs Syndrome: scoring criteria for leg movements recorded during the suggested immobilization test. Sleep Med. 2001 Jul;2(4):317-321. doi: 10.1016/s1389-9457(00)00072-1. PMID 11438248
- [Derived] Gorantla S, Ravisankar A, Trotti LM. Magnesium citrate monotherapy improves restless legs syndrome symptoms and multiple suggested immobilization test scores in an open-label pilot study. J Clin Sleep Med. 2024 Aug 1;20(8):1357-1361. doi: 10.5664/jcsm.11206. PMID 38738598
- See also: Manual used for scoring sleep and associated events — https://aasm.org/clinical-resources/scoring-manual/